CLINICAL TRIAL: NCT03562546
Title: The Effect of Structured Exercise on Chronic Venous Insufficiency: A Feasibility Trial
Brief Title: The Effect of Structured Exercise on Chronic Venous Insufficiency
Acronym: CVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shannon Hernon (Other)
Collaborators: Galway Clinic (Network)
Responsible Party: Sponsor-Investigator, Shannon Hernon, PhD Researcher, National University of Ireland, Galway, Ireland
Organization: National University of Ireland, Galway, Ireland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 369921
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Venous Insufficiency
Keywords: CVI; Calf Muscle Pump Function; Structured Exercise; Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Structured Resistance Exercise (Experimental): 12 week at home structured resistance exercise programme ('Strength From Within') using resistance bands. Under the supervision of an experienced exercise specialist.
  Interventions: Other: Strength From Within

INTERVENTIONS:
Other: Strength From Within — A 12 week at home structured resistance exercise programme using resistance bands. Participants will also receive a walking programme, a warm up and cool down, and ankle range of motion exercises.

SUMMARY:
Individuals with Chronic Venous Insufficiency (CVI) face a number of complications, such as, muscular dysfunction, limited ankle range of motion(ROM) and diminished calf muscle pump function. Exercise therapy has been shown to improve calf muscle pump function and symptoms and may provide additional therapeutic benefits. It has been reported that structured exercise has the ability to improve ankle joint range of motion, calf muscle strength and calf muscle pump function.

Participants will receive the 12-week structured resistance exercise programme, 'Strength from Within', a warm up and cool down, walking programme and range of motion exercises. Participants will complete the Short Form quality of life (SF-36) Health Survey and the venous clinical severity score questionnaire.

Baseline testing will be conducted. The following measures will be employed in the study through a baseline testing and repeated at the end of the study period (week 12): Functional ambulatory measurements, physical activity measurements (muscle endurance), isokinetic testing (strength), duplex ultrasound scanning.

A combination of upper and lower body structured exercise as well as, ankle join range of motion and a walking regimen has the potential to have a significant impact on an individual's calf muscle pump function and avoid these potentially harmful side effects of lower body exercise programmes

DETAILED DESCRIPTION:
There will be a total of sixty participants recruited for the study, with an anticipation of 40 to complete the study. Participants will complete the Physical Activity Readiness Questionnaire (PAR-Q) to ensure that they are able to participate in the structured exercise programme. If the participants' answers "yes" to any question on the Physical Activity Readiness Questionnaire (PAR-Q), he/she is ineligible to participate. Participants will also read a participant information leaflet and sign an informed consent before participating in the study. Baseline demographic will be collected at the start of the study. Participants will complete the SF-36 Health Survey at session one and session 2 (week 12). Baseline testing will be conducted. The following measures will be employed in the study through a baseline testing and repeated at the end of the study period (week 12): Functional ambulatory measurements, physical activity measurements, isokinetic testing, duplex ultrasound screening.

Upon completing baseline testing participants will have the warm-up, cool-down, stretches, all exercise demonstrated and explained to them. Participants will go through each exercise with the principal investigator to ensure understanding. The principal investigator will then describe each section of the "Strength From Within" Booklet. At the end of the first session the participants will be administered their at home structured exercise booklet, recording booklet, resistance band, warm-up and cool-down information sheet and their ankle range of motion information sheet.

The baseline meeting and the week 12 meeting will take roughly 90 minutes to complete all baseline measurements, questionnaires, isokinetic testing and demonstrations. Isokinetic testing will take a total of 32 minutes with resting periods included in the time, baseline measurements including the muscle strength and functional ambulatory measurements will take a duration of 10.5 minutes, demonstration of the home structured exercise programme will take up to 20 minutes, both questionnaires will take 5-minutes total and time left for any other questions or concerns. Extra time will be given at any point during both meetings if needed by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic venous insufficiency and a Comprehensive Classification System for Chronic Venous Disorder (CEAP) Score of 2,3,4.

Exclusion Criteria:

* Younger than 18 years
* Painful Ulceration
* Severe Cardiac Condition
* Cardiorespiratory Disease
* Failure of Physical Activity Readiness form
* American College of Sports Medicine (ACSM) Risk Classification: Class C or above
* CEAP classification of 5 or 6
* Severe mobility impairment
* Severe imbalance
* Women who are pregnant
* Women who are breastfeeding
* Those who lack capacity to consent
* Those for whom English is not the first language and have difficulty understanding written and/or spoken English
* Diagnosis of diabetes
* Diagnosis of peripheral arterial disease
* Diagnosis of peripheral neuropathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Calf Muscle Pump Function | 12 Weeks
  Duplex Ultrasound Scanning-to determine the nature and extent of venous reflux
Calf Muscle Strength | 12 Weeks
  Isokinetic Testing- Biodex
Venous Clinical Severity Score | 12 Weeks
  Questionnaire assessing severity of the patients' chronic venous insufficiency and to monitor any progression made

SECONDARY OUTCOMES:
Ankle Joint Range of Motion | 12 Weeks
  Goniometer
Overall physical strength | 12 Weeks
  Muscle Strength Endurance Testing
Quality of life | 12 Weeks
  SF-36 Short Form Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Micheál Newell, PhD, Principal Investigator — National University of Ireland, Galway, Ireland
Locations (1):
- Galway Clinic, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] O'Donovan K, Bajd T, Grace P, O'Keeffe D, Lyons G. Preliminary Evaluation of Recommended Airline Exercises for Optimal Calf Muscle Pump Activity. EJVES Extra. 2006;12(1):1-5. doi:10.1016/j.ejvsextra.2006.04.001
- [Background] Dua A, Heller JA. Advanced Chronic Venous Insufficiency. Vasc Endovascular Surg. 2017 Jan;51(1):12-16. doi: 10.1177/1538574416682175. Epub 2016 Dec 26. PMID 28024458
- [Background] White-Chu EF, Conner-Kerr TA. Overview of guidelines for the prevention and treatment of venous leg ulcers: a US perspective. J Multidiscip Healthc. 2014 Feb 11;7:111-7. doi: 10.2147/JMDH.S38616. eCollection 2014. PMID 24596466
- [Background] Brand FN, Dannenberg AL, Abbott RD, Kannel WB. The epidemiology of varicose veins: the Framingham Study. Am J Prev Med. 1988 Mar-Apr;4(2):96-101. PMID 3395496
- [Background] Callam MJ. Epidemiology of varicose veins. Br J Surg. 1994 Feb;81(2):167-73. doi: 10.1002/bjs.1800810204. PMID 8156326
- [Background] Chiesa R, Marone EM, Limoni C, Volonte M, Petrini O. Chronic venous disorders: correlation between visible signs, symptoms, and presence of functional disease. J Vasc Surg. 2007 Aug;46(2):322-30. doi: 10.1016/j.jvs.2007.04.030. Epub 2007 Jun 27. PMID 17600668
- [Background] Scott TE, LaMorte WW, Gorin DR, Menzoian JO. Risk factors for chronic venous insufficiency: a dual case-control study. J Vasc Surg. 1995 Nov;22(5):622-8. doi: 10.1016/s0741-5214(95)70050-1. PMID 7494366
- [Background] Fowkes FG, Lee AJ, Evans CJ, Allan PL, Bradbury AW, Ruckley CV. Lifestyle risk factors for lower limb venous reflux in the general population: Edinburgh Vein Study. Int J Epidemiol. 2001 Aug;30(4):846-52. doi: 10.1093/ije/30.4.846. PMID 11511615
- [Background] Sadick NS. Predisposing factors of varicose and telangiectatic leg veins. J Dermatol Surg Oncol. 1992 Oct;18(10):883-6. doi: 10.1111/j.1524-4725.1992.tb02921.x. PMID 1430543
- [Background] Iannuzzi A, Panico S, Ciardullo AV, Bellati C, Cioffi V, Iannuzzo G, Celentano E, Berrino F, Rubba P. Varicose veins of the lower limbs and venous capacitance in postmenopausal women: relationship with obesity. J Vasc Surg. 2002 Nov;36(5):965-8. doi: 10.1067/mva.2002.128315. PMID 12422106
- [Background] Evans CJ, Fowkes FG, Hajivassiliou CA, Harper DR, Ruckley CV. Epidemiology of varicose veins. A review. Int Angiol. 1994 Sep;13(3):263-70. PMID 7822904
- [Background] Browse NL. The etiology of venous ulceration. World J Surg. 1986 Dec;10(6):938-43. doi: 10.1007/BF01658644. No abstract available. PMID 3798942
- [Background] Browse N, Burnand K. CAUSE OF VENOUS ULCERATION. The Lancet. 1982;320(8304):932. doi:10.1016/s0140-6736(82)90901-1.
- [Background] Darvall KA, Sam RC, Adam DJ, Silverman SH, Fegan CD, Bradbury AW. Higher prevalence of thrombophilia in patients with varicose veins and venous ulcers than controls. J Vasc Surg. 2009 May;49(5):1235-41. doi: 10.1016/j.jvs.2008.12.017. PMID 19307088
- [Background] Allison MA, Cushman M, Callas PW, Denenberg JO, Jensky NE, Criqui MH. Adipokines are associated with lower extremity venous disease: the San Diego population study. J Thromb Haemost. 2010 Sep;8(9):1912-8. doi: 10.1111/j.1538-7836.2010.03941.x. PMID 20546124
- [Background] Serra R, Buffone G, de Franciscis A, Mastrangelo D, Molinari V, Montemurro R, de Franciscis S. A genetic study of chronic venous insufficiency. Ann Vasc Surg. 2012 Jul;26(5):636-42. doi: 10.1016/j.avsg.2011.11.036. PMID 22664280
- [Background] Anwar MA, Georgiadis KA, Shalhoub J, Lim CS, Gohel MS, Davies AH. A review of familial, genetic, and congenital aspects of primary varicose vein disease. Circ Cardiovasc Genet. 2012 Aug 1;5(4):460-6. doi: 10.1161/CIRCGENETICS.112.963439. No abstract available. PMID 22896013
- [Background] Vlajinac HD, Radak DJ, Marinkovic JM, Maksimovic MZ. Risk factors for chronic venous disease. Phlebology. 2012 Dec;27(8):416-22. doi: 10.1258/phleb.2011.011091. Epub 2012 Feb 16. PMID 22345329
- [Background] Vlajinac HD, Marinkovic JM, Maksimovic MZ, Matic PA, Radak DJ. Body mass index and primary chronic venous disease--a cross-sectional study. Eur J Vasc Endovasc Surg. 2013 Mar;45(3):293-8. doi: 10.1016/j.ejvs.2012.12.011. Epub 2013 Jan 20. PMID 23337196
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] O'Donnell TF Jr, Passman MA, Marston WA, Ennis WJ, Dalsing M, Kistner RL, Lurie F, Henke PK, Gloviczki ML, Eklof BG, Stoughton J, Raju S, Shortell CK, Raffetto JD, Partsch H, Pounds LC, Cummings ME, Gillespie DL, McLafferty RB, Murad MH, Wakefield TW, Gloviczki P; Society for Vascular Surgery; American Venous Forum. Management of venous leg ulcers: clinical practice guidelines of the Society for Vascular Surgery (R) and the American Venous Forum. J Vasc Surg. 2014 Aug;60(2 Suppl):3S-59S. doi: 10.1016/j.jvs.2014.04.049. Epub 2014 Jun 25. No abstract available. PMID 24974070
- [Background] Padberg FT Jr, Johnston MV, Sisto SA. Structured exercise improves calf muscle pump function in chronic venous insufficiency: a randomized trial. J Vasc Surg. 2004 Jan;39(1):79-87. doi: 10.1016/j.jvs.2003.09.036. PMID 14718821
- [Background] Eklof B, Perrin M, Delis KT, Rutherford RB, Gloviczki P; American Venous Forum; European Venous Forum; International Union of Phlebology; American College of Phlebology; International Union of Angiology. Updated terminology of chronic venous disorders: the VEIN-TERM transatlantic interdisciplinary consensus document. J Vasc Surg. 2009 Feb;49(2):498-501. doi: 10.1016/j.jvs.2008.09.014. PMID 19216970
- [Background] Caggiati A, Bergan JJ, Gloviczki P, Jantet G, Wendell-Smith CP, Partsch H; International Interdisciplinary Consensus Committee on Venous Anatomical Terminology. Nomenclature of the veins of the lower limbs: an international interdisciplinary consensus statement. J Vasc Surg. 2002 Aug;36(2):416-22. doi: 10.1067/mva.2002.125847. PMID 12170230
- [Background] Caggiati A, Bergan JJ, Gloviczki P, Eklof B, Allegra C, Partsch H; International Interdisciplinary Consensus Committee on Venous Anatomical Terminology. Nomenclature of the veins of the lower limb: extensions, refinements, and clinical application. J Vasc Surg. 2005 Apr;41(4):719-24. doi: 10.1016/j.jvs.2005.01.018. PMID 15874941
- [Background] Eklof B, Rutherford RB, Bergan JJ, Carpentier PH, Gloviczki P, Kistner RL, Meissner MH, Moneta GL, Myers K, Padberg FT, Perrin M, Ruckley CV, Smith PC, Wakefield TW; American Venous Forum International Ad Hoc Committee for Revision of the CEAP Classification. Revision of the CEAP classification for chronic venous disorders: consensus statement. J Vasc Surg. 2004 Dec;40(6):1248-52. doi: 10.1016/j.jvs.2004.09.027. PMID 15622385
- [Background] CRANLEY JJ, KRAUSE RJ, STRASSER ES. Chronic venous insufficiency of the lower extremity. Surgery. 1961 Jan;49:48-58. No abstract available. PMID 13696275
- [Background] Ercan S, Cetin C, Yavuz T, Demir HM, Atalay YB. Effects of isokinetic calf muscle exercise program on muscle strength and venous function in patients with chronic venous insufficiency. Phlebology. 2018 May;33(4):261-266. doi: 10.1177/0268355517695401. Epub 2017 Mar 7. PMID 28954574
- [Background] Andersen H. Reliability of isokinetic measurements of ankle dorsal and plantar flexors in normal subjects and in patients with peripheral neuropathy. Arch Phys Med Rehabil. 1996 Mar;77(3):265-8. doi: 10.1016/s0003-9993(96)90109-4. PMID 8600869
- [Background] Dix FP, Brooke R, McCollum CN. Venous disease is associated with an impaired range of ankle movement. Eur J Vasc Endovasc Surg. 2003 Jun;25(6):556-61. doi: 10.1053/ejvs.2002.1885. PMID 12787699
- [Background] Clarke Moloney M, Lyons GM, Breen P, Burke PE, Grace PA. Haemodynamic study examining the response of venous blood flow to electrical stimulation of the gastrocnemius muscle in patients with chronic venous disease. Eur J Vasc Endovasc Surg. 2006 Mar;31(3):300-5. doi: 10.1016/j.ejvs.2005.08.003. Epub 2005 Oct 20. PMID 16242978
- [Background] Boyle M, Galway B, McLaughlin T et al. Evidence-Based Clinical Protocols: 3) Anterior Cruciate Ligament Injury & Reconstruction. New York; 2006:3-3. Available at: http://www.biodex.com/sites/default/files/900521anterior.pdf.
- [Background] Boyle M, Jacoby S, McLaughlin T et al. Evidence-Based Clinical Protocols 5) Lateral Ankle Sprains. New York; 2006:5-9. Available at: http://www.biodex.com/sites/default/files/900521lateral.pdf.
- [Background] Get walking with this 12-week walking schedule - Mayo Clinic. Mayo Clinic. 2017. Available at: http://www.mayoclinic.org/healthy-lifestyle/fitness/in-depth/walking/art-20050972.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03562546/Prot_SAP_ICF_000.pdf